CLINICAL TRIAL: NCT04976868
Title: Observational Study to Evaluate the Actual Use of Elidel® in Chinese Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: Medicine Meda Pharmaceutical Information Consultancy (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: 3328
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pimecrolimus Cream 1% - Elidel®: Elidel® as prescribed within routine clinical practice
  Interventions: Drug: Pimecrolimus 1% Top Cream

INTERVENTIONS:
Drug: Pimecrolimus 1% Top Cream — Elidel® as prescribed within routine clinical practice

SUMMARY:
The primary objective of the present multicentre, prospective, non-interventional study (NIS) is gathering knowledge on the actual use and effectiveness of Elidel® in Chinese patients with mild to moderate AD affecting sensitive skin areas in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chinese ethnicity
* Patients at least 2 years old
* Signed informed consent from patient and if applicable from parent(s) or legal guardian(s) in compliance with local requirements
* Patients with mild to moderate AD and depending on the age:
* Patients 2-12 years must have:

  - SCORAD Index < 50
* Patients 13 years and older must have:

  * Affecting sensitive skin areas (e.g. face, intertriginous sites, anogenital area)
  * SCORAD Index < 50 and IGA in sensitive skin areas ≤ 3

Exclusion Criteria:

* Patients for whom Elidel® is not recommended accordingly to the Package Insert
* Patients with severe atopic dermatitis (SCORAD Index ≥ 50 or IGA in sensitive skin > 3)
* Receiving systemic glucocorticoids, antibiotics, antifungals, immunomodulators, inhibitors, antihistamines and ultraviolet radiation therapy within the last 4 weeks before inclusion;
* Receiving any topical AD-effective drugs within the last 2 weeks before inclusion;
* Pregnant and/or breastfeeding women
* Patients or parent(s) / legal guardian (as applicable) that are not able to fulfil study requirements according to physician's opinion
* Patients or parent(s) / legal guardian (as applicable) that refuse to participate to the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients at least 2 years old with mild to moderate atopic dermatitis affecting sensitive skin areas
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
SCORAD | The study ends after the Maintenance Period of at least 3 months allowing certain flexibility to respond to the routine practice. End of Study will be approx. 6 months after the inclusion depending length of the Elidel® Treatment Period.
  The primary outcome measure is the "change from baseline in SCORAD INDEX". The achievable score in SCORAD INDEX range from 0 to 103. The classification of severity would be as follows mild (<25), moderate (25-50) and severe (≥50).

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing children's Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Children's Hospital Capital Institute of Pediatrics, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Children's hospital of Chongqing medical university, Chongqing
  - The third affiliated hospital, sun yat-sen university, Guangzhou
  - The first Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Tongji Medical College Huazhong University of Science & Technology, Wuhan